CLINICAL TRIAL: NCT01395654
Title: Different Reintroduction Regimens of Antituberculosis Drugs After Development of Hepatitis During Anti-tuberculosis Treatment
Brief Title: Reintroduction Regimens After Hepatitis During Anti-tuberculosis Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201010025M
Record Dates: First submitted 2011-07-05; First posted 2011-07-15 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-11

CONDITIONS: Hepatitis; Tuberculosis, Pulmonary
MeSH Terms: conditions — Hepatitis; Tuberculosis, Pulmonary | interventions — Isoniazid; Rifampin; Pyrazinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Standard rechallenge, Slow rechallenge (Experimental)
  Interventions: Drug: isoniazid, rifampin, pyrazinamide

INTERVENTIONS:
Drug: isoniazid, rifampin, pyrazinamide — rechallenge of isoniazid (INH), rifampin (RIF), and pyrazinamide (PZA) aftr recovery from hepatitis
  Other Names: INH; RIF; PZA

SUMMARY:
Despite the availability of effective anti-tuberculosis agents that exist to treat this illness, hepatotoxicity during first-line drugs anti-tuberculosis medications (ATT) such as isoniazid (INH), rifampin (RIF), and pyrazinamide (PZA) is not uncommon and limit their use. There is no consensus on method of the reintroduction of anti-TB medications. The risk of reintroducing of a anti-TB medications could be hazardous. There are several differences between the guidelines from the ATS, BTS and the Task Force of the European Respiratory Society, the WHO and the International Union Against Tuberculosis and Lung Disease about the methods of reintroducing of anti-TB medications.

The investigators plan to do a prospective study to evaluate the outcome and safety of reintroduction of anti-TB medications after resolution of hepatitis during anti-TB treatment among TB patients in the investigators hospital.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains a leading health problem in both developing and developed countries. Despite the availability of effective chemotherapeutic agents that exist to treat this illness, hepatotoxicity during first-line drugs anti-tuberculosis medications (ATT) such as isoniazid (INH), rifampin (RIF), and pyrazinamide (PZA) is not uncommon and limit their use. In the case of confirmed moderate or severe drug-induced hepatotoxicity, treatment should be interrupted and reintroduced after the hepatotoxicity has resolved.

There is no consensus on method of the reintroduction of anti-TB medications. The risk of reintroducing of a anti-TB medications could be hazardous. There are several differences between the guidelines from the ATS, BTS and the Task Force of the European Respiratory Society, the WHO and the International Union Against Tuberculosis and Lung Disease about the methods of reintroducing of anti-TB medications.

We plan to do a prospective study to evaluate the outcome and safety of reintroduction of anti-TB medications after resolution of hepatitis during anti-TB treatment among TB patients in our hospital.

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis during anti-tuberculosis treatment
* Hold RMP, INH and PZA after hepatitis
* Age >= 18 years old
* HIV(-)
* T-bilirubin < 2.5 mg/dL
* No allergy to RMP, INH and PZA

Exclusion Criteria:

* Liver cirrhosis, child B or C
* Pregnancy and breast feeding
* Life expectation < 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The duration needed for successfully rechallenge anti-tuberculosis treatment | participants will be followed for the duration of hospital stay, an expected average of 5 weeks

SECONDARY OUTCOMES:
Number of participants with recurrence of hepatitis | participants will be followed for the duration of hospital stay, an expected average of 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jann-Yuan Wang, Principal Investigator — National Taiwan University
Locations (2):
- Taiwan (2):
  - Chest Hospital, Tainan
  - National Taiwan University Hospital, Taipei